CLINICAL TRIAL: NCT00669253
Title: Randomized Controlled Trial to Evaluate the Efficacy of Er:YAG Laser and Surgical Therapy in Treatment of Chronic Periodontitis
Brief Title: Treatment of Periodontitis Using Er:YAG Laser vs. Conventional Treatment Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/189
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Lasers, Solid-State; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Scaling and root planing at baseline and surgery for remaining deep pockets after 6 months both using Er:YAG laser
  Interventions: Procedure: Er: YAG Laser
- 2 (Active Comparator): Scaling and root planing at baseline and surgery for remaining deep pockets after 6 months both using conventional methods (ultrasonic and manual means)
  Interventions: Procedure: Conventional treatment 1(ultrasonic and manual means)
- 3 (Active Comparator): Surgery at baseline for all deep pockets using conventional methods (ultrasonic and manual means)
  Interventions: Procedure: Conventional treatment 2 (ultrasonic and manual means)

INTERVENTIONS:
Procedure: Er: YAG Laser — Scaling and root planing at baseline and surgery for remaining deep pockets after 6 months both using Er:YAG laser
  Arms: 1
Procedure: Conventional treatment 1(ultrasonic and manual means) — Scaling and root planing at baseline and surgery for remaining deep pockets after 6 months both using conventional methods : ultrasonic and manual means
  Arms: 2
Procedure: Conventional treatment 2 (ultrasonic and manual means) — Surgery at baseline for all deep pockets using conventional methods: ultrasonic and manual means
  Arms: 3

SUMMARY:
Conventional non-surgical periodontal treatment, that is, root debridement using manual and ultrasonic means at baseline and surgery using the same means after 6 months in case of persistent deep pockets (Group 1)/ Er:YAG laser used in a non-surgical approach at baseline and surgery using the same laser after 6 months in case of persistent deep pockets (Group 2)/ Surgery at baseline using manual and ultrasonic means (Group 3). All patients will undergo supragingival maintenance on a yearly basis.

ELIGIBILITY:
Inclusion Criteria:

* at least 35 years of age
* at least 18 teeth present that can be retained by means of therapy among which 4 multirooted teeth or more(wisdom teeth excluded)
* presence of at least one deep pocket per quadrant (6 mm PPD or more) with radiographic evidence of bone loss (>= 30% of root length)

Exclusion Criteria:

* pregnancy
* removable prosthesis

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth, Clinical attachment level and microbiological analysis | At baseline, 3, 6, 12, 24, 36, 48 and 60 months

SECONDARY OUTCOMES:
Gingivitis index, plaque index, bleeding on probing at the same time intervals + the number of interventions | After 5 years
Consumed time per treatment/ Patient satisfaction/comfort ( Oral Health impact Profile : OHIP )/ The estimated financial costs based on average data delivered for instance by the Belgian Society of Periodontology | After 5 years
Adverse effects described by the patient (number of painkillers taken, visual analogue scale to monitor post-operative pain, tooth sensitivity) | After 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, MD, Phd, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be